CLINICAL TRIAL: NCT06873425
Title: A Study on the Safety and Effectiveness of Limosilactobacillus Fermentum LF61 in Improving Intestinal and Immune Functions
Brief Title: Research on the Improvement of Intestinal and Immune Functions by Probiotics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK20250303
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Intestinal Health
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): Intervention with Limosilactobacillus fermentum LF61 (30 billion CFU/ day, 3g) was administered daily for 8 weeks.
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Every day to give 3 g maltodextrin intervention for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Dietary supplement: Probiotics. The trial period of this study lasts for 2 months (8 weeks), during which each participant will have 3 visits (at month 0, month 1, and month 2).
  Arms: Probiotic group
Dietary Supplement: Placebo — Dietary supplement: Placebo. The trial period of this study lasts for 2 months (8 weeks), during which each participant will have 3 visits (at month 0, month 1, and month 2).
  Arms: Placebo group

SUMMARY:
Evaluate the effectiveness and safety of Limosilactobacillus fermentum LF61 as a food supplement compared to a placebo in improving intestinal and immune functions in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to undergo 3 follow-up visits during the intervention period
2. Be willing to provide blood, urine and stool samples 2 times during the intervention period
3. Willing to self-administer one of the 7 probiotics (BI45, BBi32, LS97, LB42, LF61, LH76, LR08)/placebo once a day during the intervention period
4. Good eyesight, can read and write, can wear glasses
5. Have good hearing and be able to hear and understand all instructions during the intervention -

Exclusion Criteria:

1. Digestive diseases, mainly gastrointestinal diseases (celiac disease, ulcerative colitis, Crohn's disease)
2. Have a serious neurological condition (epilepsy, stroke, severe head trauma, meningitis in the last 10 years, brain surgery, brain tumor, prolonged coma - not including general anaesthesia)
3. Have received/are receiving treatment for the following mental disorders: alcohol/drug/substance abuse dependence, schizophrenia, psychosis, bipolar disorder
4. Take medication for depression or low mood
5. Internal organ failure (heart, liver or kidney failure, etc.)
6. Have received radiation or chemotherapy in the past
7. have undergone a general anesthesia procedure/procedure within the past three years, or plan to undergo a general anesthesia procedure/procedure within the next 3 months during this trial period
8. Have had hepatitis (hepatitis B, hepatitis C), HIV or syphilis in the past -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of concentration of antimicrobial peptide LL-37 | Week 0 and Week 8
  Detected by Enzyme-Linked Immunosorbent Assay (ELISA).
Change in calcarein concentration | Week 0 and Week 8
  Detected by Enzyme-Linked Immunosorbent Assay (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- Xu fei, Zhengzhou, Henan, China